CLINICAL TRIAL: NCT06250504
Title: Long-acting HIV Pre-Exposure Prophylaxis Integrated With Community-based Sexual and Reproductive Health in South Africa (LAPIS): A Hybrid (1a) Cluster Randomised Controlled Phase 3B Trial of Effectiveness and Implementation
Brief Title: Long-Acting HIV Pre-Exposure Prophylaxis Integrated With Sexual and Reproductive Health - cRCT
Acronym: LAPIS
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Africa Health Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: cRCT-PrEP-AC-001
Record Dates: First submitted 2023-12-15; First posted 2024-02-09 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections | interventions — cabotegravir; Dapivirine; Contraceptive Devices, Female; Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination; Tenofovir; dolutegravir

STUDY DESIGN:
Intervention Model Description: A hybrid phase 3B effectiveness implementation type 1a cluster randomised control trial (cRCT)
Who Masked: Investigator, Outcomes Assessor
Masking Description: The statistician and clinical team will not participate in the public randomisation. The statistician will remain blinded until the analysis plan has been finalised and the database is locked. Investigators remain blinded to allocation throughout. The participants and intervention delivery teams are not blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention: Choice of long-acting PrEP and PEP added to Thetha Nami ngithethe nawe (Experimental): Tailored peer-led psychosocial support and social mobilisation into community based SRH and differentiated HIV care and prevention, including a choice of effective PrEP or PEP.
  At the mobile AYFS in the intervention clusters nurses will offer the choice of either daily oral tenofovir/emtricitabine or injectable long acting cabotegravir (CAB LA) to be delivered to adolescents and young adults at risk of HIV acquisition. Those who decline will have the option of three monthly dapivarine vaginal rings or Post Exposure Prophylaxis (PEP) packs (tenofovir/lamuvidine/dolutegravir) to take home.
  Peer navigators will promote long-acting PrEP in addition to oral PrEP. As part of the peer mentorship package, the peer naviators will remind young people of their follow-up visits.
  Interventions: Drug: APRETUDE (cabotegravir) 600 mg\3 mL; Drug: DAPIRING (Dapivirine) 25mg Vaginal Ring; Drug: tenofovir disoproxil and emtricitabine; Drug: Tenofovir Disoproxil, Lamuvidine and Dolutegravir
- Control (Enhanced SoC): Thetha Nami ngithethe nawe (Active Comparator): Tailored peer-led psychosocial support and social mobilisation into community based SRH and differentiated HIV care and prevention, including oral tenofovir/emtricitabine PrEP.
  In the mobile AYFS, young people are offered self-taken vaginal swabs or urine testing for sexually transmitted infections (STIs), family planning support and syndromic and aetiological management for STIs; HIV counselling and two POCT; immediate initiation of ART if living with HIV and oral tenofovir/emtricitabine PrEP if HIV test is negative and they are suitable.
  Peer navigators in control clusters will promote oral PrEP during their community based health promotion activities. As part of the peer mentorship package, the peer naviators will remind young people of their follow-up visits and if required accompany young people to the mobile clinics.
  Interventions: Drug: tenofovir disoproxil and emtricitabine

INTERVENTIONS:
Drug: APRETUDE (cabotegravir) 600 mg\3 mL — choice of 2-monthly injectable long acting cabotegravir. The initial visit will be followed by planned visit for the first injection, one month visit for second injection, and then 2-monthly CAB LA injections with repeat HIV testing and pregnancy testing, and referral to peer navigators for adherence and retention support. We will conduct HIV testing, STI testing, Hep B, Hep C, and safety bloods (Full Blood Count, Creatinine, Liver Function Tests) at baseline, HIV testing two monthly, and annual safety bloods, alongside annual STI testing.
  Arms: Intervention: Choice of long-acting PrEP and PEP added to Thetha Nami ngithethe nawe
Drug: DAPIRING (Dapivirine) 25mg Vaginal Ring — The initial visit is followed by a 7-day phone call, 3-monthly follow-up. Each follow-up will include repeat HIV testing (POCT x2 and dry blood spots for HIV ELISA) and pregnancy testing, syndromic management of STIs, and referral to peer navigators for adherence support and PrEP/ART and if applicable contraception refills. Safely bloods (full blood count, creatinine, liver function tests) will follow national guidelines. Currently we aim to do baseline and annual safety bloods, alongside annual STI testing
  Arms: Intervention: Choice of long-acting PrEP and PEP added to Thetha Nami ngithethe nawe
Drug: tenofovir disoproxil and emtricitabine — The initial visit is followed by a 7-day phone call, 3-monthly follow-up. Each follow-up will include repeat HIV testing (POCT x2 and dry blood spots for HIV ELISA) and pregnancy testing, syndromic management of STIs, and referral to peer navigators for adherence support and PrEP/ART and if applicable contraception refills. Safely bloods (full blood count, creatinine, liver function tests) will follow national guidelines. Currently we aim to do baseline and annual safety bloods, alongside annual STI testing
Drug: Tenofovir Disoproxil, Lamuvidine and Dolutegravir — The initial visit is followed by a 7-day phone call, 3-monthly follow-up. Each follow-up will include repeat HIV testing (POCT x2 and dry blood spots for HIV ELISA) and pregnancy testing, syndromic management of STIs, and referral to peer navigators for adherence support and PrEP/ART and if applicable contraception refills. Safely bloods (full blood count, creatinine, liver function tests) will follow national guidelines. Currently we aim to do baseline and annual safety bloods, alongside annual STI testing
  Arms: Intervention: Choice of long-acting PrEP and PEP added to Thetha Nami ngithethe nawe

SUMMARY:
The goal of this hybrid (1a) Cluster Randomised Controlled Trial phase 3B trial is to evaluate the effectiveness and implementation of offering a choice of HIV Pre-Exposure Products (PrEP) through community-based sexual and reproductive health services, on PrEP uptake and retention, and population prevalence of sexually transmissible HIV amongst adolescents and young adults living in rural South Africa.

Researchers will compare adding the choice of long-acting PrEP, i.e. two monthly injectable cabotegravir (CAB LA) or dapiravine vaginal ring and HIV post exposure prophylaxis packs to daily oral PrEP integrated with community-based SRH in the 20 intervention clusters with standard of care (SoC), daily oral PrEP integrated with community-based SRH in the 20 control clusters, on uptake and retention on PrEP. We hypothesise that offering a choice of long-acting or oral PrEP and PEP within the community-based delivery of SRH services will overcome the challenges and barriers to effective use of oral daily PrEP and lead to a population-level effect on uptake and retention on PrEP and thus the prevalence of sexually transmissible HIV amongst 15-30 year olds living in rural KwaZulu-Natal, South Africa.

DETAILED DESCRIPTION:
This is a pragmatic trial of adding in a choice of South African Health Products Registration Authority (SAHPRA) approved newer PrEP products - APRETUDE (cabotegravir) 600 mg\3 mL: DAPIRING (Dapivirine) 25mg Vaginal Ring:56/20.2.8/0979 (22/11/2022) - to the current national department of health approved oral daily PrEP with TVF/FTC (Tenofovir disoproxil/emtricitabine), Objective 1. To measure the effectiveness of the choice of oral and long-acting PrEP, including injectable (CAB LA) and vaginal ring (DapiRing), and post exposure prophylaxis (PEP) on increasing effective uptake (adoption), retention, and adherence of PrEP compared to oral PrEP in young people aged 15-30 in rural South Africa and to estimate the preliminary effect on transmissible HIV and HIV incidence.

Objective 2. To understand real-world implementation:

2.1 To explore the acceptability, appropriateness, preference, and reach of CABLA from the perspective of young people aged 15-30 and their communities in rural South Africa 2.2 To understand the feasibility, affordability, and scalability of delivering CABLA through community-based PrEP with SRH.

2.3 To identify implementation challenges and practical solutions for CABLA initiation, laboratory monitoring (e.g. RNA testing), and safe stopping within nurse-led and rural community-based clinical settings 2.4 To evaluate the safety and tolerability of CABLA compared to oral PrEP

ELIGIBILITY:
Inclusion Criteria:

All young men and women aged 15-30 who are residing in the 40 administrative clusters in the study district and attend any integrated SRH/HIV service

Documented HIV negative test

Suitable for PrEP and/or already on PrEP

Weight > 35 kg

Understand the required dosing schedule and HIV testing.

Aware that details can be shared with a peer navigator to support their follow-up

If pregnant or breast feeding and/or planning to become pregnant participant can be offered CAB LA, if risk of acquiring HIV out weighs unknown risk of CAB LA, but must understand that safety in pregnancy or breast feeding for CAB LA has not been established and oral daily PrEP is a safe alternative.

Exclusion Criteria:

History or presence of allergy to the study drugs or their components

Investigator assessment find them not suitable

Additional exclusion criteria for specific products:

CAB LA: Taking medication that is contraindicated (Carbamazepine, oxcarbazepine, phenobarbital, phenytoin, Rifampin, rifapentine) and Severe mental health disorder, Hep B surface antigen positive, living with hepatitis C and not yet treated, or abnormal liver function tests (ALT more than two times the upper limit of normal)

DapiRing: Pregnancy.

Ages: 15 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes
Enrollment: 2000 (Estimated)
Dates: Start 2024-02-27 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Uptake PrEP | This will be evaluated among participants aged 16-30 years in the cross-sectional surveys at 14 months
  Defined as the proportion of young people who have taken up any PrEP (oral, injectable, ring, or PEP).
Retention on PrEP | This will be measured in the clinical cohort of consenting clinic attendeeswho start or are on PrEP/PEP during the first 10 months of the trial.
  Defined as attending at least one follow-up appointment after PrEP/PEP initiation, including for HIV testing.

SECONDARY OUTCOMES:
The prevalence of transmissible HIV. | 14 months
  We will measure this outcome as the proportion of those living with HIV and have a detectable HIV viral load, defined as having an HIV viral load of >= 400 copies per ml, during our final survey round.
Uptake of risk informed HIV prevention | 14 months
  Defined as the proportion of 16-30 year olds who are aware of their HIV status and have undergone a HIV risk assessment to inform HIV prevention and/or are on/start HIV treatment if living with HIV.
PrEP Reach (Adoption) | 14 months
  Proportion of those at greatest risk adopting (taking up) PrEP or PEP in each arm. Greatest risk is defined as an aggregate exposure disaggregated by gender that includes any of the following factors: out of school (aged <= 18) or unemployed (aged >18) and/or engaged in transactional sex or sex work and/or harmful alcohol use (AUDIT scale) and/or experience physical, sexual or emotional violence (validated tool) and/or food poverty (recent experience of hunger)
PrEP delivery cost and cost-effectiveness | 14 months
  cost per effective PrEP uptake in each arm
Adverse events | 14 months
  Proportion discontinue or switch due to adverse events in each arm
Proportion of men and women aged 16-30 at risk of acquiring HIV or transmitting HIV | 14 months
  If living with HIV (a detectable viral load + condomless sex + not on ART), or, if not living with HIV (condomless sex + not on PrEP)

OTHER OUTCOMES:
Sexual and reproductive health | 14 months
  uptake of family planning, teenage pregnancies and sexually transmitted infection prevalence in each arm
Improved socioeconomic outcomes | 14 months
  Defined as proportion in school (aged <= 18) or unemployed (aged >18) and/or food secure (no recent experience of hunger) in each arm.
improved mental health | 14 months
  Proportion with PHQ9 score consistent with common mental disorder in each arm

CONTACTS AND LOCATIONS:
Locations (1):
- Africa Health Research Institute, Somkele, KwaZulu-Natal, South Africa

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: After the primary analysis has been completed and publicaly shared

REFERENCES:
- [Derived] Busang J, Zuma T, Chimbindi N, Ngoma N, Herbst C, Okesola N, Dreyer J, Smit T, Bird K, Mtolo L, Behuhuma N, Lebina L, Hendrickson C, Miot J, Hanekom W, Herbst K, Seeley J, Copas A, Baisley K, Shahmanesh M; LAPIS Study Team. Long-acting HIV pre-exposure prophylaxis integrated with community-based sexual and reproductive health services in South Africa (LAPIS): study protocol for a hybrid (1a) cluster randomised controlled phase 3B trial of effectiveness and implementation. BMC Public Health. 2026 Jan 20. doi: 10.1186/s12889-025-24889-1. Online ahead of print. PMID 41559582